CLINICAL TRIAL: NCT00812877
Title: Mineral Trioxide Aggregate (MTA) vs. Calcium Hydroxide (CaOH) in Direct Pulp Capping in NW PRECEDENT (Northwest Practice-based REsearch Collaborative in Evidence-based DENTistry Practices.
Brief Title: Pulp Capping With Two Different Agents
Acronym: MTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: University of Washington (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Thomas J. Hilton, DMD, MS, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDCR-16752; U01DE016750 (NIH)
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Dental Pulp Exposure
Keywords: pulp capping; MTA; CaOH; Mineral Trioxide Aggregate; Calcium Hydroxide
MeSH Terms: conditions — Dental Pulp Exposure | interventions — mineral trioxide aggregate; Pemetrexed; Calcium Hydroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mineral Trioxide Aggregate (Active Comparator): Pulp capping agent, Mineral Trioxide Aggregate used as a direct pulp cap
  Interventions: Drug: Mineral Trioxide Aggregate
- Calcium Hydroxide (Active Comparator): Pulp capping agent, Calcium Hydroxide used as a direct pulp cap
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Drug: Mineral Trioxide Aggregate — Pulp capping agent, Mineral TrioxideAggregate
  Other Names: MTA
  Arms: Mineral Trioxide Aggregate
Drug: Calcium Hydroxide — Pulp capping agent, Calcium Hydroxide
  Arms: Calcium Hydroxide

SUMMARY:
The purpose of this study is to determine if MTA or calcium hydroxide are more effective as pulp capping agents

DETAILED DESCRIPTION:
The purpose of this study was to test two dental products used as direct pulp capping agent for the permanent teeth. The two products were mineral trioxide aggregate and calcium hydroxide.

A direct pulp capping consists of covering an exposed tooth pulp (the inside portion of the tooth where the blood vessels and nerve supply the tooth) with a medication to maintain tooth vitality. Different events can cause the pulp to be exposed, for example a deep cavity, or an accident where the outer portion of the tooth fractures. When this occurs, it is sometimes possible to place a medicine over the top of the exposure (a "cap") in an effort to allow the pulp to heal on its own. Our study intended to compare two of those medicines, calcium hydroxide and mineral trioxide aggregate, both Federal Drug Administration (FDA) approved products, to determine if one performed better than the other.

The study was conducted with patients recruited by Northwest PRECEDENT practitioners. The practitioners interested in participating in the study were randomized (assigned by chance) to one of the two intervention groups: a treatment group (mineral trioxide aggregate) and a control group (calcium hydroxide).

Direct pulp capping was completed on permanent (adult) teeth with pulps exposed due to decay, trauma (injury) or mechanical exposure. Treated teeth were followed over two years to determine how well they responded to the treatment.

All patients who had a pulp exposure of a permanent tooth were eligible for the study. These patients were further asked to participate in the study if they satisfied the inclusion criteria for the study and did not present any of the exclusion criteria stated in the study protocol.

A tooth that received a pulp cap was treated in the following manner: After a tooth pulp had been exposed and the tooth was found to be suitable for a pulp cap, the exposure and surrounding area was cleaned by gentle rinsing with water. A cotton pellet moistened with 5.25% sodium hypochlorite was placed over the exposure and allowed to sit for 1-2 minutes. This procedure was used to control pulp bleeding and remove the germs from that area. After the initial period, the cotton pellet was removed and the area inspected. If bleeding continued, a new cotton pellet moistened in the sodium hypochlorite solution was reapplied to the area for an additional several minutes. This was repeated until bleeding was controlled or the practitioner decided that pulp capping was not appropriate for the situation. Once the bleeding was controlled from the exposure, one of the two pulp capping agents was applied to the pulp exposure site.

Practices were assigned by chance into one of two treatment groups, those that completed direct pulp capping with mineral trioxide aggregate and those that completed direct pulp capping with calcium hydroxide, both FDA approved agents for this purpose. The handling characteristics of the two materials were so different, that it was not practical to blind the practitioners as to which material they were using. Likewise, training in the use of each material was required. It was believed that it was more important that the practitioner become familiar and competent in the use of one of the materials to ensure it was used appropriately, than it was to have practitioners use both materials and confuse procedures between them. Since time was a critical element in the success or failure of direct pulp capping, the patients were consented to participate in the study after the procedure was done. A resin-modified glass ionomer liner (e.g. Vitrebond, Fuji Lining Cement, Fuji II LC, Vitremer) was placed over the pulp capping agent. This liner sealed the pulp capping agent and protected the pulp from being infiltrated with bacteria. After the resin-modified glass ionomer lining material was set, the final filling was placed.

Two types of instruments were used in this study:

Study participant data collection form This form collected two types of data: demographic and clinical data. The demographic part gathered information regarding patient age, gender, and race. The clinical form collected data regarding the clinical and x-ray evaluation of the tooth treated with a direct pulp cap: condition of the tooth, the type of pulp exposure (by decay, by injury or during tooth preparation), patients' complaints regarding the tooth, and results of diagnostic tests (x-ray, pain to biting or temperature, etc) were recorded.

Practitioner feedback survey A survey was administered to all practitioners who participated in the study. This survey included a series of questions designed to evaluate the communication between the member practitioners and the network, practitioner/staff training, patient recruitment, obtaining informed consent, data collection and data transmission, including the electronic data capture system. The survey also tried to determine how well the offices were able to combine the research in a regular daily office schedule in order to determine if a research project would affect the normal day-to-day routine.

The intent of this study was to find out which of the two products yielded better results as a pulp capping agent. In order to detect this, the failure rates in the two treatment groups were compared using statistical tests. Distributions of covariates in the two treatment groups were compared and clinical judgment was used to identify covariates with serious group imbalances that would cause an unusual result for the primary analysis. Logistic regression was used to compare failure rates while adjusting for any covariates that were imbalanced between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient 7 years old or older who requires a direct pulp cap of a permanent tooth.
2. The tooth must exhibit a vital pulp upon exposure.
3. The exposure can be due to mechanical, traumatic or carious causes.
4. Patient will be available for the two year follow-up period.

Exclusion Criteria:

1. Any primary tooth requiring a direct pulp cap.
2. Tooth demonstrates any radicular radiolucency on a radiograph.
3. Tooth exhibits spontaneous pain.
4. Tooth exhibits lingering (more than 5 seconds) pain to temperature or biting stimulus.
5. Non-English and/or non-Spanish speaking subjects.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hilton, DMD, MS, Principal Investigator — NW PRECEDENT
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Hilton TJ. Keys to clinical success with pulp capping: a review of the literature. Oper Dent. 2009 Sep-Oct;34(5):615-25. doi: 10.2341/09-132-0. No abstract available. PMID 19830978
- [Result] Hilton TJ, Ferracane JL, Mancl L; Northwest Practice-based Research Collaborative in Evidence-based Dentistry (NWP). Comparison of CaOH with MTA for direct pulp capping: a PBRN randomized clinical trial. J Dent Res. 2013 Jul;92(7 Suppl):16S-22S. doi: 10.1177/0022034513484336. Epub 2013 May 20. PMID 23690353

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-five dental practices recruited and enrolled subjects between May 2009 and March 2011.
Pre-assignment Details: Randomization was done on a practice level rather than a patient level. The handling characteristics of the two materials were so dissimilar that it was not feasible to blind the practitioners as to which material they were using.
Period: Overall Study
Arm/Group | Mineral Trioxide Aggregate | Calcium Hydroxide
Started | 195 | 181
Completed | 158 | 130
Not Completed | 37 | 51

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mineral Trioxide Aggregate | Calcium Hydroxide | Total
Number analyzed (Participants) | 195 | 181 | 376
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34 | 31 | 65
  Between 18 and 65 years | 147 | 138 | 285
  >=65 years | 14 | 12 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (18.6) | 36.3 (18.0) | 37.5 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 94 | 191
  Male | 98 | 87 | 185
Region of Enrollment [Number; unit: participants]
  United States | 195 | 181 | 376

OUTCOME MEASURES:

1. Primary Outcome: Tooth Survival
Description: No recommendation for tooth extraction or root canal therapy. Only one tooth was enrolled/assessed per participant.
Time Frame: Up to two years
Population: 12 subjects were excluded in the Mineral Trioxide Aggregate group due to lack of follow-up (4 subjects were non-responsive; unable to contact 6 subjects; 2 subjects changed dentists) and 6 subjects were in the Calcium Hydroxide group (2 subjects were non-responsive; unable to contact 3 subjects; 1 subject was incarcerated).
Measure: Number; unit: participants
Arm/Group | Mineral Trioxide Aggregate | Calcium Hydroxide
Number analyzed (Participants) | 183 | 175
participants | 158 | 130
Statistical Analysis 1: Comparison: Mineral Trioxide Aggregate vs Calcium Hydroxide; Test type: Superiority or Other; p = .046, Log Rank — A clustered permutation test with 10,000 random permutations based on the log rank test statistic was used for the primary treatment comparison to account for censoring and to ensure proper test size given the number of practices; Hazard Ratio (HR) = 2.35, 95% CI 2-sided [1.19 to 4.66] — A confirmatory analysis, adjusted for patient, dentist, and tooth characteristics, and follow-up time, was performed using marginal proportional hazards regression with robust standard error estimates accounting for clustering by practice

2. Secondary Outcome: Pulp Vitality
Description: No evidence of pulpal resorption or calcification or periradicular radiolucency
Time Frame: Up to two years
Measure: Number; unit: participants
Arm/Group | Mineral Trioxide Aggregate | Calcium Hydroxide
Number analyzed (Participants) | 183 | 175
participants | 155 | 130

ADVERSE EVENTS:
Arm/Group | Mineral Trioxide Aggregate | Calcium Hydroxide
Serious Adverse Events (participants affected / at risk) | 2/195 | 1/181
Other Adverse Events (participants affected / at risk) | 5/195 | 2/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mineral Trioxide Aggregate (N=195) | Calcium Hydroxide (N=181)
Death of patient (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Ovarian cancer
Death of Patient (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Lung cancer
Death of patient (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pulmonary embolism
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mineral Trioxide Aggregate (N=195) | Calcium Hydroxide (N=181)
Not feeling well (General disorders) | 1 (1) | 0 (0) — Possibly nausea due to pain medication.
H1N1 flu (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cough and fever
Toothache on non-study tooth (Infections and infestations) | 3 (3) | 0 (0) — Carious tooth
Temperature sensitivity and dull ache in upper left quadrant (Infections and infestations) | 0 (0) | 1 (1) — Probably related to caries in study tooth
Diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Diagnosed while participating in study

LIMITATIONS AND CAVEATS:
1. Randomization was by practice therefore, some dentists may have used a material with which they had little familiarity.
2. Lack of on-going monitoring of study procedures may have caused an inordinate number of failures in one practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No